CLINICAL TRIAL: NCT05337150
Title: Evaluating a Remotely Delivered Behavioral Weight Loss Intervention Using an Ad Libitum Plant-Based Diet Versus a Balanced Calorie Deficit Diet
Brief Title: Remotely Delivered Behavioral Weight Loss Using an Ad Libitum Plant-Based Diet Versus a Balanced Calorie Deficit Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HEALTHQUEST
Record Dates: First submitted 2022-03-25; First posted 2022-04-20 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-01

CONDITIONS: Obesity; Overweight
Keywords: vegetarian; behavioral weight loss; weight loss; dietary self-monitoring; obesity
MeSH Terms: conditions — Obesity; Overweight; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle Modification with a Balanced Calorie Deficit Diet (Experimental): Lifestyle modification intervention with a balanced calorie deficit diet (i.e., participants will be prescribed a calorie goal and will track their dietary intake in order to meet this goal).
  Interventions: Behavioral: Lifestyle Modification Intervention; Behavioral: Balanced Calorie Deficit Eating Plan
- Lifestyle Modification with an Ad Libitum Whole Food Plant-Based Eating Plan (Experimental): Lifestyle modification intervention with an ad libitum whole food plant-based diet (i.e., participants will eat, ad libitum, fruits, vegetables, starches, legumes, and whole grains, and will avoid eating processed foods, refined oils, and animal products)
  Interventions: Behavioral: Lifestyle Modification Intervention; Behavioral: Ad Libitum Whole Food Plant-Based Eating Plan

INTERVENTIONS:
Behavioral: Lifestyle Modification Intervention — For the first 12-weeks of the study, participants will complete weekly web modules in which they will learn cognitive-behavioral strategies to support lifestyle modification. Participants will also receive weekly phone coaching calls for the first 12-weeks of the study, and monthly coaching calls thereafter for the remainder of the 24-week study period.
Behavioral: Balanced Calorie Deficit Eating Plan — Participants will be prescribed a calorie target between 1200 and 1800 depending upon baseline weight and personal preference. Participants will be asked to monitor their dietary intake using MyFitnessPal and to submit food logs weekly. Calorie reduction content will be based primarily on the Diabetes Prevention Program protocol and adapted from existing behavioral treatment protocols. Individuals will receive general guidelines on eating a healthy diet, including reducing saturated fat, processed foods, refined sugars, and refined carbohydrates, and increasing intake of lean proteins, whole grains, and fruits and vegetables, but will be encouraged to flexibly decide which areas of their diet to modify to reduce calorie intake.
  Arms: Lifestyle Modification with a Balanced Calorie Deficit Diet
Behavioral: Ad Libitum Whole Food Plant-Based Eating Plan — Participants will be prescribed a whole food plant-based (WFPB) low-fat vegan diet promoting intake of fruits, vegetables, starches, legumes, and whole grains. Participants will be encouraged to avoid processed foods, refined oils, and animal products (meat, fish, eggs, and dairy products), and to minimize consumption of high-fat plant-based foods. An adapted traffic-light diet chart will outline foods to eat daily, limit, and avoid. Participants will be advised to eat until satiation and not restrict energy intake. Participants will be asked to consume 50 μg vitamin B12 (methylcobalamin) daily. WFPB nutrition counseling content will be based upon existing successful programs. Each week, participants will complete a simplified dietary self-monitoring food frequency questionnaire aligned to correspond with the traffic light diet chart.
  Arms: Lifestyle Modification with an Ad Libitum Whole Food Plant-Based Eating Plan

SUMMARY:
This pilot randomized controlled trial will compare a remotely delivered behavioral weight loss program with a balanced calorie deficit diet (the current gold-standard) to a behavioral weight loss program with an ad libitum whole food plant-based diet (WFPBD) amongst adults with overweight/obesity (N = 52). The 6-month intervention will consist of 3 months of moderate-intensity intervention (weekly online modules and brief coaching calls), then a low-intensity period (3 calls over 3-months). Assessments will occur at baseline, 6-weeks, 12-weeks, and post-treatment (6-months). Acceptability, dietary adherence, weight, quality of life, depressive symptoms, and subjective appetite will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* BMI 27-50 kg/m2
* Ages 18-75 years
* Resides in the U.S.
* Consistent access to internet at home
* Proficient skill level in speaking, writing, and understanding English
* Reporting a desire to lose weight
* Consistently available for 15-minute once-weekly video appointment between the hours of 8 AM and 7 PM EST
* Willing to follow a whole food plant-based diet or a traditional calorie-reduced diet for the study duration
* Individuals must provide consent for the research team to contact their personal physician if necessary, to provide clearance or to consult about rapid weight loss

Exclusion Criteria:

* Currently pregnant or breastfeeding or planned pregnancy within the study period
* Recent weight loss (≥ 5% weight loss in 3-months prior to the study)
* History of bariatric surgery
* Currently following a low-fat plant-based diet
* Medical condition (e.g., cancer, type I diabetes, renal failure), current substance use problem, or psychiatric condition (e.g., active substance abuse, eating disorder) that may pose a risk to the participant during intervention or cause a change in weight
* Recently began or changed the dose of a medication that can cause significant change in weight
* Planning on quitting cigarette smoking over the program period
* Participation in a concurrent weight loss program during the study period
* Medical diagnosis currently influencing weight or appetite
* Medical condition that would limit ability to participate in this program (for example, mild stroke, diabetes if taking insulin, head trauma, cognitive disorder)
* Acute suicidality
* Currently meets criteria for regular loss-of-control eating (i.e., ≥ 9 binge episodes in past 3 months
* Currently reports engaging in a compensatory behavior

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2022-05-29 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-03-24 (Actual)

PRIMARY OUTCOMES:
Weight Change | Measured at each assessment baseline, mid-treatment (6- and 12-weeks) and post-treatment (6-months).
  Weight loss will be self-reported by participants using a standardized weighing procedure. Participants will weigh themselves in lightweight clothes without shoes with a digital scale accurate to 0.1 kg. Percent weight loss at 6-months will be calculated as the percentage loss in initial body weight at baseline by the time of the post-treatment assessment.

SECONDARY OUTCOMES:
Subjective Appetite as assessed by visual analogue scale (VAS) | Measured at baseline, mid-treatment (6- and 12-weeks) and post-treatment (6-months).
  Subjective appetite will be assessed using 6 visual analogue scale items (VAS) inquiring about past-week hunger, fullness, the degree to which hunger made it difficult to follow the prescribed diet, preoccupation with thoughts of food, and being bothered by hunger on a visual analogue scale of 0-100. Scores on the fullness item will be reversed, such that higher scores will indicate greater subjective appetite.

OTHER OUTCOMES:
Dietary adherence as assessed by food frequency questionnaire (FFQ) | Measured at baseline, mid-treatment (6- and 12-weeks) and post-treatment (6-months).
  Dietary adherence in the whole food plant-based diet (WFPBD) condition will be assessed with an adapted 7-item food frequency questionnaire (FFQ). Each day for 7 days, participants will indicate whether they ate each of the "green zone" food categories (veggies/fruits, leafy greens, whole gains/starches, beans/lentils), whether they ate less than 3 servings of "yellow zone" foods, the "red-zone" foods consumed (and servings of). To evaluate whether intake of green/yellow/red-zone foods changes more in the WFPBD condition than in the balanced calorie deficit diet (BCDD) condition, those in the BCDD condition will complete the FFQ at each assessment point. To evaluate dietary adherence in the BCDD condition, calorie-tracking adherence will be examined. Dietary adherence on a given day will be defined as the overall number of days participants tracked at least two eating occasions.
Quality of Life Change as assessed by the 36-item Short-Form General Health Survey (SF-36) | Measured at baseline, mid-treatment (12-weeks) and post-treatment (6-months).
  Quality of life will be assessed using the 36-item Short-Form General Health Survey (SF-36; Ware, Kosinski, & Keller, 1994; Ware & Sherbourne, 1992), which assesses eight domains: physical functioning, limits due to physical health, pain, general health, energy/fatigue, social functioning, emotional wellbeing, and mental health. Scores will be converted to a 0 to 100 scale, with higher scores indicating better functioning. This scale produces both physical health (PH) and mental health (MH) component summaries.
Intentions to continue adhering to dietary prescription as assessed by a Future Intentions Questionnaire | Measured at post-treatment (12-weeks and 6-months).
  Intentions to continue adhering to dietary prescription will be assessed with a 3-item self-report measure ("Future Intentions Questionnaire"). On a Likert scale ranging from 1 (Not at all) to 5 (Completely), participants will respond to face-valid questions asking about plans to continue adhering to the prescribed program diet (sample item: "I plan to follow the diet from this program moving forward") and the feasibility of the program diet (sample item: "The diet in this program is straightforward to follow moving forward"). Accompanying the measure, participants will receive a brief reminder of their dietary prescription (i.e., the traffic light diet chart in the whole food plant-based diet condition, or the calorie goal and daily calorie tracking requirement in the balanced calorie deficit diet condition). Items will be averaged to create a measure of intentions to adhere to the prescribed diet; higher scores indicate greater adherence.
Depressive Symptoms as assessed by the Beck Depression Inventory-II (BDI-II) | Measured at baseline, mid-treatment (6- and 12-weeks) and post-treatment (6-months).
  To assess depressive symptoms, the Beck Depression Inventory-II (BDI-II; Dozois et al., 1998) will be administered-a 21-item measure of somatic (e.g., appetite), affective (e.g., sadness) and cognitive (e.g., self-criticalness) dimensions of depressive symptomology. Participants will indicate how they have been feeling during the past week and make responses on a Likert scale ranging from 0 (e.g., I don't cry any more than I used to) to 3 (e.g., I feel like crying but I can't), with higher scores indicating greater levels of depressive symptoms.
Program acceptability as assessed by a program acceptability questionnaire | Measured at post-treatment (6-months).
  Overall program acceptability will be assessed post-treatment with a questionnaire adapted from prior work (Bradley et al., 2017) that will ask participants to report how satisfied they were with the program, the degree to which they found the program helpful, and the likelihood they would recommend it to family or friends using a Likert scale ranging from 1 (Not at all) to 5 (Very much). Scores will be averaged across conditions to create mean program acceptability scores. Higher scores will indicate greater program acceptability.
Dietary acceptability as assessed by a diet acceptability questionnaire | Measured at post-treatment (6-months).
  Participants will indicate the degree to which they found their diet to be acceptable by indicating, on a Likert scale, how difficult they found the diet to follow (1-Very Easy - 5-Very difficult) with regards to: following the diet as a whole, cooking, dietary tracking, staying full, and managing cravings. Participants will also indicate how time-consuming they found their diet (1-Not at all time-consuming - 5-Very time-consuming), and how confident they felt in their ability to follow their diet (1-Not at all - 5-Very much so). Scores will be averaged across items to create mean dietary acceptability scores.
Association between social support vs. social sabotage (as assessed by Ball & Crawford) at Week 12 (mid-treatment) and percent weight loss at 6-months (post-treatment). | Measured at mid-treatment (12-weeks) and post-treatment (6-months).
  To assess social support vs. social sabotage, participants will complete the Social Support and Sabotage Scale from Ball & Crawford (2006). On this measure, participants separately rate the degree to which friends and family act in ways that support or hinder their healthy eating efforts with a Likert scale ranging from 1 (Almost never) to 5 (Almost always). Scores will be averaged for each subscale to compute: 1) support for health behaviors from friends, 2) support for health behaviors from family, 3) sabotage for health behaviors from friends, and 4) sabotage for health behaviors from family.
Fatigue as assessed by the FACIT Fatigue | Measured at baseline, mid-treatment (6- and 12-weeks) and post-treatment (6-months).
  Self-reported fatigue will be measured using the Functional Assessment of Chronic Illness Therapy - Fatigue Scale (FACIT Fatigue), a 13-item self-report questionnaire that assesses level of fatigue during an individual's usual daily activities over the past week on a Likert scale ranging from 4 (not at all fatigued) to 0 (very much fatigued) (Webster et al., 2003). Scores will be reversed such that higher scores indicate greater levels of fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Evan Forman, PhD, Principal Investigator — Drexel University
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No